CLINICAL TRIAL: NCT00618228
Title: A Single Dose, Two-Period, Two-Treatment, Randomized Crossover Bioequivalency Study of 750 mg Balsalazide Capsules Under Fasting Conditions
Brief Title: Bioequivalency Study of Balsalazide Capsules Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst/Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BALS-02
Record Dates: First submitted 2008-01-30; First posted 2008-02-19 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — balsalazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Balsalazide

SUMMARY:
The objective of this study was to assess bioequivalence of a potential generic 750 mg balsalazide disodium capsule formulation compared with Salix Pharmaceutical's 750 mg balsalazide disodium capsule, Colazal, following a single 750 mg dose, under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant finding on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enyzme altering drugs.
* History of allergic or adverse response to balsalazide, mesalamine, salicylates, or other related drugs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2004-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, 7 day washout

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D>, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceuticals Research Services, Houston, Texas, United States